CLINICAL TRIAL: NCT06857955
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, 12 Months Treatment Duration, Dose Finding Study, to Evaluate Efficacy, Safety and Pharmacodynamics of QCZ484 in Mild to Moderate Hypertensive Patients
Brief Title: A Study to Identify an Optimal Dose of QCZ484 in Mild to Moderate Hypertensive Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CQCZ484A12201
Record Dates: First submitted 2025-03-03; First posted 2025-03-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: QCZ484; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo Control (Placebo Comparator): Placebo
  Interventions: Other: Saline
- QCZ484 Dose 1 (Experimental): QCZ484 Dose 1 solution for injection
  Interventions: Drug: QCZ484
- QCZ484 Dose 2 (Experimental): QCZ484 Dose 2 solution for injection
  Interventions: Drug: QCZ484
- QCZ484 Dose 3 (Experimental): QCZ484 Dose 3 solution for injection
  Interventions: Drug: QCZ484
- QCZ484 Dose 4 (Experimental): QCZ484 Dose 4 solution for injection
  Interventions: Drug: QCZ484
- QCZ484 Dose 5 (Experimental): QCZ484 Dose 5 solution for injection
  Interventions: Drug: QCZ484

INTERVENTIONS:
Other: Saline — 0.9% sodium chloride saline solution
  Arms: Placebo Control
Drug: QCZ484 — Solution of Injection
  Arms: QCZ484 Dose 1; QCZ484 Dose 2; QCZ484 Dose 3; QCZ484 Dose 4; QCZ484 Dose 5

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of QCZ484 or placebo, given subcutaneously, every 6 months, at different dose levels in patients with mild to moderate hypertension

DETAILED DESCRIPTION:
Phase 2b, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy, safety, and pharmacodynamics of QCZ484 with mild to moderate hypertension (HTN). Multiple doses of QCZ484 will be tested against placebo, administered as subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Males or females aged 18 to 75 years.
3. Diagnosis of hypertension.
4. Hypertension treatment naive or on maximum 2 anti-HTN medications and able to undergo washout for 4 weeks.
5. Mean sitting SBP ≥140 mmHg measured by OBPM and mean 24 hr SBP ≥130 mmHg and <160 mmHg measured by ABPM.
6. Participants able to understand and comply with study procedures.

Exclusion Criteria:

1. Known history of secondary hypertension.
2. Orthostatic hypotension.
3. Laboratory parameter assessments outside of range at screening.
4. Evidence of hepatic disease.
5. Medical condition, other than hypertension, requiring treatment with RAAS inhibitor.
6. Any history of congestive heart failure.
7. Current or history of intolerance to ACEi and/or ARBs.
8. Clinically significant cardiac arrhythmias, high-grade AV block and third-degree AV block within 6 months prior to screening.
9. Acute myocardial infarction (AMI) or unstable angina, or any percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within 12 months prior to screening. Any history of ischemic or hemorrhagic stroke or transient ischemic attack any time prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2028-04-05 (Estimated)

PRIMARY OUTCOMES:
Change in Mean 24hr SBP by ABPM | Baseline, Month 3
  Change from baseline at Month 3 in mean 24hr systolic blood pressure (SBP) by ambulatory blood pressure measurement (ABPM)

SECONDARY OUTCOMES:
Change in Mean 24hr SBP by ABPM | Baseline, Month 6
  Change from baseline at Month 6 in mean 24hr SBP by ABPM
Change in SBP by OBPM | Baseline, Month 3 and 6
  Change from baseline at Month 3 and 6 in SBP by office blood pressure measurement (OBPM)
Participants achieving SBP<130 mmHg or SBP reduced by ≥10 mmHg by ABPM | Baseline, Month 3 and 6
  Proportion of responders defined as participants achieving SBP<130 mmHg or SBP reduced by ≥10 mmHg from baseline, at Month 3 and 6 by ABPM
Change in DBP by ABPM and OBPM | Baseline, Month 3 and 6
  Change from baseline at Month 3 and 6 on diastolic blood pressure (DBP) by ABPM and OBPM
Number of participants with AEs | Up to Month 18
  Number of participants with AEs by treatment group, including changes in vital signs and laboratory results qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (76):
- United States (71):
  - SEC Clinical Research LLC, Andalusia, Alabama
  - UAB St Vincents, Birmingham, Alabama
  - Longwood Research, Huntsville, Alabama
  - The Center for Clinical Trials, Saraland, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - NICRs Research Center, Garden Grove, California
  - Valiance Clinical Research, Huntington Park, California
  - Downtown L.A. Research Center Inc, Los Angeles, California
  - Clinical Trials Research Sacramento, Sacramento, California
  - Encompass Clinical Research, Spring Valley, California
  - Clinical Research of Brandon LLC, Brandon, Florida
  - ALL Medical Research LLC, Cooper City, Florida
  - National Research Institute, Hialeah, Florida
  - Cen Exel RCA, Hollywood, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Entrust Clinical Research, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - American Research Centers of FL, Pembroke Pines, Florida
  - Cen Exel FCR, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Centricity Research, Columbus, Georgia
  - Javara Research, Fayetteville, Georgia
  - Velocity Clinical Research, Savannah, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Cedar Crosse Research Ct, Chicago, Illinois
  - Eagle Clinical Research, Chicago, Illinois
  - Synexus Clinical Research US, Evansville, Indiana
  - Velocity Clin Research Sioux City, Sioux City, Iowa
  - Alliance for Multispecialty Research, Wichita, Kansas
  - Velocity Clinical Res Baton Rouge, Baton Rouge, Louisiana
  - Southern Clin Research Clinic, Zachary, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - AA Medical Research Center, Flint, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Synexus Clinical Research US Inc, Richfield, Minnesota
  - David M Headley Clinic, Port Gibson, Mississippi
  - Healthcare Research Network II LLC, Hazelwood, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Clin Rsrch Consult a JCCT Company, Kansas City, Missouri
  - Velocity Clin at Pioneer Heart Inst, Lincoln, Nebraska
  - AMR Las Vegas, Las Vegas, Nevada
  - CenExel HRI, Berlin, New Jersey
  - Velocity Clinical Research, Binghamton, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Accellacare of Rocky Mount, Rocky Mount, North Carolina
  - Accellacare of Salisbury, Salisbury, North Carolina
  - CR Services Acquisition US, Columbus, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Velocity Clinical Research Medford, Medford, Oregon
  - TCV Clinical Studies, Linwood, Pennsylvania
  - Velocity Clinical Research, Union, South Carolina
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee
  - Velocity Clinical Research Austin, Austin, Texas
  - North Hills Medical Research Inc, Bedford, Texas
  - Synergy Group Medical LLC, Houston, Texas
  - Biopharma Informatic, Katy, Texas
  - Synergy Groups Medical LLC, Missouri City, Texas
  - Sun Research Institute, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - AMR Layton, Layton, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Centricity Research Suffolk Fam Med, Suffolk, Virginia
  - MultiCare Ins Research Innovation, Puyallup, Washington
  - Velocity Clinical Research Spokane, Spokane, Washington
- Japan (4):
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Novartis is commited to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.